CLINICAL TRIAL: NCT05587192
Title: Radical Prostatectomy Without Prostate Biopsy Following 18F-PSMA-1007 PET/CT Based on a Diagnostic Model: a Single-center, Single-arm, Open-label Study
Brief Title: Radical Prostatectomy Without Prostate Biopsy Following PSMA PET/CT Based on Diagnostic Model
Acronym: RPWPB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, TaoTao, Associate professor, Associate chief physician, Anhui Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNOTOB
Record Dates: First submitted 2022-10-17; First posted 2022-10-19 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; PSMA-1007; PET-CT; Biopsy; prostate-specific antigen; mpMRI; Diagnosis
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-PSMA-1007 PET/CT based on USTC diagnostic model (Experimental): Patinets will complete the 18F-PSMA-1007 PET/CT based USTC diagnostic model firstly. If clinically significant prostate cancer is considered by 18F-PSMA-1007 PET/CT. Patinets will receive radical prostatectomy directly or undergo prostate biopsy according to patients own decisions, patients with negative results in prostate biopsy will be asked to complete rebiopsy after 3 months.
  Interventions: Diagnostic Test: 18F-PSMA-1007 PET/CT based on diagnostic model

INTERVENTIONS:
Diagnostic Test: 18F-PSMA-1007 PET/CT based on diagnostic model — All enrolled patients will receive 18F-PSMA-1007 PET/CT based USTC diagnostic model before gaining the final pathological diagnosis to be used as experimental arm.

SUMMARY:
The goal of this prospective, single-center, single-arm trial is to evaluate the positive predictive values between 18F-PSMA-1007 PET/CT based on diagnostic model in patients with suspicious of prostate cancer. The main question and our aim to answer is:

• Can these patients with clinically significant prostate cancer in 18F-PSMA-1007 PET/CT based on diagnostic model undergo radical prostatectomy directly without prostate biopsy.

Participants will be asked to accomplish the test of serum PSA, mpMRI, then, the eligible patients (The probability of the diagnostic model to predict clinically significant prostate cancer was greater than or equal to 60 percent) need perform 18F-PSMA-1007 PET/CT. Finally, patients will receive radical prostatectomy directly if prostate cancer is considered by 18F-PSMA-1007 PET/CT.

DETAILED DESCRIPTION:
Study Design and Setting SNOTOB study is a prospective, single-center, single-arm and open-label clinical study and conducted in the First Affiliated Hospital of USTC in China. Patients who have no surgical contraindications and meet the enrollment criteria will be recruited to the study. Subsequently, we will recommend these patients to accept radical prostatectomy without prostate biopsy directly. Before the operation, patients and their family member will be fully informed of the surgical risks, the necessity to perform a prostate biopsy for pathologic confirmation, the possibility of benign prostatic disease and the other alternative therapeutic methods including active surveillance, radiotherapy, and focal therapies and so on. Finally, the diagnostic performance of our noninvasive diagnostic strategy will be verified with the pathological results.

Screening and Enrollment The noninvasive diagnostic strategy in this study consists of a prostate cancer diagnostic model and 18F-prostate-specific membrane antigen-1007 positron emission tomography/computed tomography (18F-PSMA-1007 PET/CT) examination in series. After the patients complete the serum prostate-specific antigen (PSA) test and multiparameter magnetic resonance imaging (mpMRI), we can obtain the information of prostate-specific antigen density (PSAD) and prostate imaging-reporting and data system version 2.1 (PI-RADS v2.1) score. Then, patients' risk probability of clinically significant prostate cancer (csPCa) will be calculated by the online diagnostic nomogram (website: https://ustcprostatecancerprediction.shinyapps.io/dynnomapp/). When the prediction probability of csPCa is equal or greater than 0.60, 18F-PSMA-1007 PET/CT will be applied for further diagnosis. If patients are still considered as csPCa after 18F-PSMA-1007 PET/CT examinations, we define this condition as positive result of our noninvasive diagnostic strategy. These patients meet our criteria of this study. Of note, patients with prediction probability less than 0.60 will no longer undergo 18F-PSMA-1007 PET/CT examinations, and patients with risk probability equal or greater than 0.60 but negative 18F-PSMA-1007 PET/CT examinations will not meet the enrollment criteria too.

ELIGIBILITY:
Inclusion Criteria:

1. Men with clinically suspected prostate cancer (abnormal DRE or PSA);
2. Complete the test of serum PSA and examination of mpMRI;
3. 4 ng/ml ≤serum total PSA<100ng/ml;
4. The probability of the diagnostic model to predict clinically significant prostate cancer was greater than or equal to 60 percent;
5. Prostate cancer is considered by 18F-PSMA-1007 PET/CT;
6. Meet the surgical indications for radical prostatectomy.

Exclusion Criteria:

1. Incomplete information of serum PSA tests or mpMRI;
2. serum total PSA<4ng/ml or ≥ 100 ng/ml;
3. The probability of the diagnostic model to predict clinically significant prostate cancer was less than 60 percent;
4. Prostate cancer is not considered by 18F-PSMA-1007 PET/CT;
5. Patients who have negative results in the previous prostate biopsy;
6. Patients refuse radical prostatectomy or still choose prostate biopsy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Detection rate of clinically significant prostate cancer | Immediately after prostatectomy
  Detection rate of clinically significant prostate cancer which defined as Gleason score ≥ 3+4.

SECONDARY OUTCOMES:
Detection rate of prostate cancer | Immediately after prostatectomy
  Detection rate of prostate cancer which defined as Gleason score ≥ 3+3.
Detection of high-grade prostate cancer | Immediately after prostatectomy
  Detection of high-grade prostate cancer which defined as Gleason score ≥ 4+3.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Tao, MD Ph.D, Study Chair — The First Affiliated Hospital of USTC
Locations (1):
- The First Affiliated Hospital of USTC, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xia C, Dong X, Li H, Cao M, Sun D, He S, Yang F, Yan X, Zhang S, Li N, Chen W. Cancer statistics in China and United States, 2022: profiles, trends, and determinants. Chin Med J (Engl). 2022 Feb 9;135(5):584-590. doi: 10.1097/CM9.0000000000002108. PMID 35143424
- [Background] Rebello RJ, Oing C, Knudsen KE, Loeb S, Johnson DC, Reiter RE, Gillessen S, Van der Kwast T, Bristow RG. Prostate cancer. Nat Rev Dis Primers. 2021 Feb 4;7(1):9. doi: 10.1038/s41572-020-00243-0. PMID 33542230
- [Background] Ilic D, Djulbegovic M, Jung JH, Hwang EC, Zhou Q, Cleves A, Agoritsas T, Dahm P. Prostate cancer screening with prostate-specific antigen (PSA) test: a systematic review and meta-analysis. BMJ. 2018 Sep 5;362:k3519. doi: 10.1136/bmj.k3519. PMID 30185521
- [Background] Mottet N, van den Bergh RCN, Briers E, Van den Broeck T, Cumberbatch MG, De Santis M, Fanti S, Fossati N, Gandaglia G, Gillessen S, Grivas N, Grummet J, Henry AM, van der Kwast TH, Lam TB, Lardas M, Liew M, Mason MD, Moris L, Oprea-Lager DE, van der Poel HG, Rouviere O, Schoots IG, Tilki D, Wiegel T, Willemse PM, Cornford P. EAU-EANM-ESTRO-ESUR-SIOG Guidelines on Prostate Cancer-2020 Update. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2021 Feb;79(2):243-262. doi: 10.1016/j.eururo.2020.09.042. Epub 2020 Nov 7. PMID 33172724
- [Background] Naji L, Randhawa H, Sohani Z, Dennis B, Lautenbach D, Kavanagh O, Bawor M, Banfield L, Profetto J. Digital Rectal Examination for Prostate Cancer Screening in Primary Care: A Systematic Review and Meta-Analysis. Ann Fam Med. 2018 Mar;16(2):149-154. doi: 10.1370/afm.2205. PMID 29531107
- [Background] Duffy MJ. Biomarkers for prostate cancer: prostate-specific antigen and beyond. Clin Chem Lab Med. 2020 Feb 25;58(3):326-339. doi: 10.1515/cclm-2019-0693. PMID 31714881
- [Background] Mazzone E, Stabile A, Pellegrino F, Basile G, Cignoli D, Cirulli GO, Sorce G, Barletta F, Scuderi S, Bravi CA, Cucchiara V, Fossati N, Gandaglia G, Montorsi F, Briganti A. Positive Predictive Value of Prostate Imaging Reporting and Data System Version 2 for the Detection of Clinically Significant Prostate Cancer: A Systematic Review and Meta-analysis. Eur Urol Oncol. 2021 Oct;4(5):697-713. doi: 10.1016/j.euo.2020.12.004. Epub 2020 Dec 25. PMID 33358543
- [Background] Sathianathen NJ, Omer A, Harriss E, Davies L, Kasivisvanathan V, Punwani S, Moore CM, Kastner C, Barrett T, Van Den Bergh RC, Eddy BA, Gleeson F, Macpherson R, Bryant RJ, Catto JWF, Murphy DG, Hamdy FC, Ahmed HU, Lamb AD. Negative Predictive Value of Multiparametric Magnetic Resonance Imaging in the Detection of Clinically Significant Prostate Cancer in the Prostate Imaging Reporting and Data System Era: A Systematic Review and Meta-analysis. Eur Urol. 2020 Sep;78(3):402-414. doi: 10.1016/j.eururo.2020.03.048. Epub 2020 May 20. PMID 32444265
- [Background] Berry B, Parry MG, Sujenthiran A, Nossiter J, Cowling TE, Aggarwal A, Cathcart P, Payne H, van der Meulen J, Clarke N. Comparison of complications after transrectal and transperineal prostate biopsy: a national population-based study. BJU Int. 2020 Jul;126(1):97-103. doi: 10.1111/bju.15039. Epub 2020 Apr 6. PMID 32124525
- [Background] Hubner N, Shariat S, Remzi M. Prostate biopsy: guidelines and evidence. Curr Opin Urol. 2018 Jul;28(4):354-359. doi: 10.1097/MOU.0000000000000510. PMID 29847523
- [Background] Tao T, Wang C, Liu W, Yuan L, Ge Q, Zhang L, He B, Wang L, Wang L, Xiang C, Wang H, Chen S, Xiao J. Construction and Validation of a Clinical Predictive Nomogram for Improving the Cancer Detection of Prostate Naive Biopsy Based on Chinese Multicenter Clinical Data. Front Oncol. 2022 Jan 21;11:811866. doi: 10.3389/fonc.2021.811866. eCollection 2021. PMID 35127526
- [Background] Neels OC, Kopka K, Liolios C, Afshar-Oromieh A. Radiolabeled PSMA Inhibitors. Cancers (Basel). 2021 Dec 13;13(24):6255. doi: 10.3390/cancers13246255. PMID 34944875
- [Background] Scheltema MJ, Chang JI, Stricker PD, van Leeuwen PJ, Nguyen QA, Ho B, Delprado W, Lee J, Thompson JE, Cusick T, Spriensma AS, Siriwardana AR, Yuen C, Kooner R, Hruby G, O'Neill G, Emmett L. Diagnostic accuracy of 68 Ga-prostate-specific membrane antigen (PSMA) positron-emission tomography (PET) and multiparametric (mp)MRI to detect intermediate-grade intra-prostatic prostate cancer using whole-mount pathology: impact of the addition of 68 Ga-PSMA PET to mpMRI. BJU Int. 2019 Nov;124 Suppl 1:42-49. doi: 10.1111/bju.14794. Epub 2019 Jul 9. PMID 31287613
- [Background] Emmett L, Buteau J, Papa N, Moon D, Thompson J, Roberts MJ, Rasiah K, Pattison DA, Yaxley J, Thomas P, Hutton AC, Agrawal S, Amin A, Blazevski A, Chalasani V, Ho B, Nguyen A, Liu V, Lee J, Sheehan-Dare G, Kooner R, Coughlin G, Chan L, Cusick T, Namdarian B, Kapoor J, Alghazo O, Woo HH, Lawrentschuk N, Murphy D, Hofman MS, Stricker P. The Additive Diagnostic Value of Prostate-specific Membrane Antigen Positron Emission Tomography Computed Tomography to Multiparametric Magnetic Resonance Imaging Triage in the Diagnosis of Prostate Cancer (PRIMARY): A Prospective Multicentre Study. Eur Urol. 2021 Dec;80(6):682-689. doi: 10.1016/j.eururo.2021.08.002. Epub 2021 Aug 28. PMID 34465492
- [Background] Meissner VH, Rauscher I, Schwamborn K, Neumann J, Miller G, Weber W, Gschwend JE, Eiber M, Heck MM. Radical Prostatectomy Without Prior Biopsy Following Multiparametric Magnetic Resonance Imaging and Prostate-specific Membrane Antigen Positron Emission Tomography. Eur Urol. 2022 Aug;82(2):156-160. doi: 10.1016/j.eururo.2021.11.019. Epub 2021 Dec 6. PMID 34887117
- [Derived] Wang C, Dong Q, Liu X, Ni M, Xie Q, Xiao J, Tao T. Protocol for SNOTOB study: radical prostatectomy without prostate biopsy following 18F-PSMA-1007 PET/CT based on a diagnostic model: a single-centre, single-arm, open-label study. BMJ Open. 2023 Nov 19;13(11):e073983. doi: 10.1136/bmjopen-2023-073983. PMID 37984956

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT05587192/Prot_SAP_001.pdf